CLINICAL TRIAL: NCT05967702
Title: A 3-year Cross-sectional Assessment of the Tianjin Child and Adolescent Large-scale Eye Study
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2023040
Record Dates: First submitted 2023-07-09; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a school-based, cross-sectional study to assess the incidence and prevalence, risk factors of myopia among schoolchildren in both eye-use environment, eye-use habits, lifestyle, and family and subjective factors before and during COVID-19. Large population and representative study subjects. Environmental exposure and daily within and out-of-school activities will be evaluated in a random subgroup.

DETAILED DESCRIPTION:
Myopia is the most common refractive error and a major reason for reducing uncorrected visual acuity among schoolchildren. It was reported that during COVID-19, home confinement resulted in a significant increase in myopia due to the changed lifestyle of schoolchildren dramatically. However, it is unclear which kind of risk factors should be the first to bear the brunt before and during COVID-19. And which factors should be emphasized and confronted as the optimum strategy for myopia prevention and control? This cohort study aims to determine the risk factors, prevalence, and incidence of myopia, and SE changes among schoolchildren before and during COVID-19, hence identifying the factors that impact the onset and progression of myopia.

This is a 3-year cross-sectional study. This study plans to enroll 126,810 participants (aged 6-18 years) from Tianjin, China. All grade students from 10 regions of Tianjin City, China will be analyzed. Over a 3-year follow-up period, students will receive detailed eye examinations annually and complete questionnaires about eye-use environment, eye-use habits, lifestyle, and family and subjective factors. In a 5% random sample size of this cohort study, outdoor activity, light intensity, eye use habits, and eye use environment data will be obtained using objective measuring devices. Myopia was defined as spherical equivalent refractive (SER) of ≤ -0.5D.

ELIGIBILITY:
Inclusion Criteria:

* All 6-18 years students

Exclusion Criteria:

* No eye diseases such as cataracts, glaucoma, keratoconus, etc.
* No psychiatric disorders
* Astigmatism ≤ -6.00D

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All 6-18-year students with no significant systemic or eye diseases are eligible for vision screening
Sampling Method: Non-Probability Sample
Enrollment: 126810 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of myopia | One day measurement
  Myopia was defined as an equivalent spherical refraction ≤ -0.50D in either eye
Prevalence of high myopia | One day measurement
  High myopia was defined as an equivalent spherical refraction ≤ -6.00D in either eye

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Director — Tianjin Eye Hospital and Eye Institute, Nankai University Affiliated Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Result] Modjtahedi BS, Abbott RL, Fong DS, Lum F, Tan D; Task Force on Myopia. Reducing the Global Burden of Myopia by Delaying the Onset of Myopia and Reducing Myopic Progression in Children: The Academy's Task Force on Myopia. Ophthalmology. 2021 Jun;128(6):816-826. doi: 10.1016/j.ophtha.2020.10.040. Epub 2020 Dec 30. PMID 33388160
- [Result] Hu Y, Zhao F, Ding X, Zhang S, Li Z, Guo Y, Feng Z, Tang X, Li Q, Guo L, Lu C, Yang X, He M. Rates of Myopia Development in Young Chinese Schoolchildren During the Outbreak of COVID-19. JAMA Ophthalmol. 2021 Oct 1;139(10):1115-1121. doi: 10.1001/jamaophthalmol.2021.3563. PMID 34529002